CLINICAL TRIAL: NCT06802939
Title: RTMS for Refractory Auditory Hallucinations Based on Personalized Targets Using Magnetoencephalography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEG-AHTM-2024
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Refractory Auditory Hallucinations; Schizophrenia
Keywords: auditory hallucinations; rTMS; MEG; Individualized targets
MeSH Terms: conditions — Hallucinations; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Exploratory self controlled clinical intervention trial. Pseudo stimulus intervention in weeks 1-2, for a total of 10 days. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical intervention for before-after study in the same patient with auditory hallucinations (Other): Pseudo stimulus intervention in weeks 1-2, for a total of 10 days. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — RTMS using pseudo stimulus intervention in weeks 1-2, for a total of 10 days. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days. Application of rTMS for 1Hz low-frequency intervention, with intervention parameters of 1400 sessions, 100% exercise threshold, and a total of 23 minutes per session. After each target intervention, rest for half an hour to one hour.

SUMMARY:
This study is an before-after study in the same patient, which enrolled 36 psychiatric patients with refractory auditory hallucinations. The target of patient intervention relies on the results of magnetoencephalography localization. The medication and dosage remain unchanged during the intervention period. The investigators assume that the intervention targets for each auditory hallucination patient are individualized.

DETAILED DESCRIPTION:
This study is divided into two parts:

1. Target determination. Firstly, MEG data of the patient's resting and task states are collected, and a precise localization model using magnetoencephalography is applied to locate the precise location of the patient's abnormal signals in the brain, which is then used as the intervention target. Based on the patient's tolerance for single day intervention, the appropriate number of targets is generally 2-4. The upper limit of targets is 4.
2. RTMS individualized intervention. Application of rTMS for 1Hz low-frequency intervention, with intervention parameters of 1400 sessions, 100% exercise threshold, and a total of 23 minutes per session. After each target intervention, rest for half an hour to one hour. The pseudo stimulation intervention lasted for 10 days in the first and second weeks, and the scale was evaluated after the end of the pseudo stimulation. After resting for 2 weeks, enter the 3-4 weeks of real stimulation, with 5 days of intervention per week for a total of 10 days. 2-4 targets per day, 23 minutes per target, with 30-60 minutes between interventions for each target. After the fourth week, evaluate the scale. Follow up evaluations will be conducted on the 7th, 14th, 30th, 60th, and 90th day after intervention. By analyzing and evaluating data, explore individualized treatment plans for auditory hallucinations in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Must be able to right-handed
* Primary school education or above
* Understand and sign a written informed consent form (jointly signed by the guardian and the participant if under 18 years old)
* Existence of persistent auditory hallucinations (defined as: taking sufficient antipsychotic medication for at least 6 months, combined with 3 antipsychotic medications still ineffective, and no significant improvement in auditory hallucinations symptoms, with an AHRS score still>12)

Exclusion Criteria:

* MECT treatment within the past 3 months
* Major physical illnesses (organic lesions such as sensory and motor disorders, neurological disorders, and traumatic brain injury)
* Taboo symptoms for rTMS treatment (such as intracranial metal implants)
* Aggressive behavior and an impulse to damage equipment
* Metal (including orthodontic treatment, dental implants) and tattoos inside the body
* Claustrophobia

Ages: 13 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction rate of the AHRS scale | From enrolment to the end of the 2-week pseudostimulation treatment. From 2 weeks rest after the end of pseudostimulation treatment to the end of 2 weeks of true stimulation treatment.
  AHRS (Auditory Hallucinations Rating Scale) is a scale used to assess patients' auditory hallucinations within the past 24 hours. The minimum score of the AHRS scale is 0, indicating the absence of auditory hallucination symptoms, while the maximum score represents the most severe level of symptoms. The specific numerical values need to refer to the version of the scale being used.

SECONDARY OUTCOMES:
Reduction rate of the PSYRATS scale | From enrolment to the end of the 2-week pseudostimulation treatment. From 2 weeks rest after the end of pseudostimulation treatment to the end of 2 weeks of true stimulation treatment.
  PSYRATS(Psychotic Symptom Rating Scales) is a scale used to assess patients' auditory hallucinations within the past week. The PSYRATS scale is a semi-structured interview scale designed for assessing the multidimensional symptoms of auditory hallucinations and delusions, consisting of 17 items. The scale is scored on a 0-4 rating scale, with detailed explanations for each rating level, and is administered by trained staff to evaluate patients. Theoretically, the minimum score of the PSYRATS scale is 0 (when all items are scored 0), while the maximum score is 68 (when all items are scored 4). A higher score indicates more severe symptoms.
Reduction rate of the PNASS scale | From enrolment to the end of the 2-week pseudostimulation treatment. From 2 weeks rest after the end of pseudostimulation treatment to the end of 2 weeks of true stimulation treatment.
  PNASS (Positive and Negative Syndrome Scale) is a scale for evaluating Psychiatric disorders. Each item is scored on a scale from 1 to 7, with 1 being the lowest score and 7 being the highest. Therefore, the minimum possible score on the PANSS is 30, and the maximum is 210. A higher score indicates more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
All research data sharing related to humans requires hospital approval.

REFERENCES:
- [Background] Lynch CJ, Elbau IG, Ng TH, Wolk D, Zhu S, Ayaz A, Power JD, Zebley B, Gunning FM, Liston C. Automated optimization of TMS coil placement for personalized functional network engagement. Neuron. 2022 Oct 19;110(20):3263-3277.e4. doi: 10.1016/j.neuron.2022.08.012. Epub 2022 Sep 15. PMID 36113473
- [Background] Cash RFH, Weigand A, Zalesky A, Siddiqi SH, Downar J, Fitzgerald PB, Fox MD. Using Brain Imaging to Improve Spatial Targeting of Transcranial Magnetic Stimulation for Depression. Biol Psychiatry. 2021 Nov 15;90(10):689-700. doi: 10.1016/j.biopsych.2020.05.033. Epub 2020 Jun 7. PMID 32800379